CLINICAL TRIAL: NCT06722612
Title: Cohort Study of Chemotherapy Combined With Targeted Adjuvant Therapy for High-risk HER2 Positive and Lymph Node Negative Early Breast Cancer
Brief Title: Chemotherapy Combined With Targeted Therapy for High-risk HER2 Positive and Lymph Node Negative Early Breast Cancer
Acronym: TaxCbHER2
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z166
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer
Keywords: Taxane; target therapy; carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taxanes combined with carboplatin: Paclitaxel drugs (paclitaxel, liposomal paclitaxel, docetaxel, albumin paclitaxel), carboplatin chemotherapy, combined with targeted therapy with trastuzumab, for a total of 6 cycles, followed by targeted therapy with trastuzumab for 1 year.
- Taxanes: Taxanes (paclitaxel, liposomal paclitaxel, docetaxel, albumin paclitaxel), combined with targeted therapy with trastuzumab and pertuzumab, for a total of 6 cycles, followed by targeted therapy with trastuzumab and pertuzumab for 1 year.

SUMMARY:
Human epidermal growth factor receptor 2 (HER2) positive breast cancer is a molecular subtype with high malignancy and easy recurrence and metastasis. The emergence of HER2 targeted drugs has greatly improved the prognosis and survival of such patients. At present, for HER2 positive breast cancer patients with negative lymph nodes, chemotherapy drugs combined with trastuzumab is the current standard treatment scheme, and in most cases, chemotherapy uses a combination of two drugs, while the main beneficiaries of the target treatment of trastuzumab and pertuzumab are concentrated in the group of patients with positive lymph nodes. Can the use of target therapy to de-escalation chemotherapy and further achieve a strategy of high efficacy and low toxicity. It is planned to explore the efficacy and safety of T1-T2, HER2 positive early breast cancer patients with negative lymph nodes to achieve chemotherapy reduction based on risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* 1) Treated in Peking University People's Hospital and underwent radical resection with hospitalization records;
* 2) Postoperative pathology confirmed invasive breast cancer, pathological staging was T2, N0, HER2 positive, and accompanied by one of the high-risk factors (G3, or hormone receptor negative);
* 3) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Preoperative neoadjuvant therapy;
* 3) Patients with metastatic breast cancer or bilateral breast cancer;
* 4) Failure to perform radical surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invasive breast cancer, pathological staging was T2, N0, HER2 positive, and accompanied by one of the high-risk factors (G3, or hormone receptor negative)
Sampling Method: Probability Sample
Enrollment: 2916 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.

SECONDARY OUTCOMES:
invasive disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
distant disease free survival | 5 years
  Time from study enrollment to distant recurrence and metastasis
breast cancer specific survival | 5 years
  Time from study enrollment to death due to breast cancer
overall survival | 5 years
  Time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China